CLINICAL TRIAL: NCT04175509
Title: Improving Post-Operative Pain and Recovery in Gynecologic Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aultman Health Foundation (Other)
Responsible Party: Principal Investigator, Michaela Beynon, Principal Investigator, Aultman Health Foundation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2019.08.20.MB
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Results first posted 2021-08-19 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Postoperative Pain; Opioid Use; Acetaminophen
Keywords: Postoperative Pain; Minimally-invasive Hysterectomy; Opioid Use; Acetaminophen; Hysterectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rectal acetaminophen (Active Comparator): Patients will receive two 650mg suppositories rectally of acetaminophen for a total dose of 1300mg at the end of surgery.
  Interventions: Drug: Rectal acetaminophen
- Intravenous acetaminophen (Active Comparator): Patients will receive one dose of 1000mg of acetaminophen, administered intravenously, at the end of surgery.
  Interventions: Drug: Intravenous acetaminophen

INTERVENTIONS:
Drug: Rectal acetaminophen — Rectal 1300mg
  Arms: Rectal acetaminophen
Drug: Intravenous acetaminophen — Intravenous 1000mg
  Arms: Intravenous acetaminophen

SUMMARY:
This is a clinical investigation to determine the efficacy of rectal versus intravenous acetaminophen in patients undergoing a minimally invasive hysterectomy. All women will receive acetaminophen either rectally or intravenously immediately postoperative, prior to extubation. Patient's will be randomly assigned to either the rectal acetaminophen or the intravenous acetaminophen group. Patient outcomes will be measured through a Numeric Rating Scale (NRS) from 0-10 for pain scores, and total opioid consumption measured in morphine milligram equivalent (MME) for the first 24 hours following surgery, or upon discharge, whichever comes first.

DETAILED DESCRIPTION:
Patient's undergoing major gynecologic surgery require effective postoperative pain management in order to enhance recovery and ultimately allow patients to return to their preoperative functional state. Traditionally, acute postoperative pain control has been achieved largely with the use of opioid medications. Excessive use of opioids can have adverse effects on the recovery process. Side effects include, but are not limited to dizziness, sedation, nausea/vomiting, respiratory depression, euphoria, constipation, and abuse. In addition, opioid monotherapy can delay post-operative ambulation, contribute to prolonged hospital stay and resumption of activities of daily living, and furthermore, have long-term sequelae for individuals as well as society at whole.

Over the past decade, a multimodal approach to pain management has been explored in attempts to optimally treat acute postoperative pain. This approach is one of the keys to improving the recovery process.

Acetaminophen is a non-opioid analgesic with a well-established safety and tolerability profile that is commonly used in multimodal approach to treating surgical pain. It is available in oral, rectal and Intravenous (IV) formulation. IV acetaminophen in particular is increasingly used for pain control after surgery as it has demonstrated a significant analgesic benefit in a variety of surgery types by reduction in pain intensity while decreasing total opioid use. Many studies have evaluated the efficacy of acetaminophen based on route of administration. A systematic review demonstrated that there is no clear indication for intravenous acetaminophen for patients who can tolerate an oral dosage as there was no difference if efficacy outcomes. This is valuable information as the cost of IV acetaminophen is exponentially more than the oral form. Although the oral form of acetaminophen is as efficient as controlling pain when compared to IV, and is notably cheaper, it is not the best option for the nauseated patient or patients whom are restricted from oral intake following surgery. Rectal acetaminophen is therefore a feasible alternative option in such patients.

Data on the use of rectal acetaminophen in adults for postoperative pain management is limited. Pettersson and colleagues (2005) compared oral, rectal and IV paracetamol in day surgery patients. Although they demonstrated significantly higher plasma paracetamol concentrations in patients who received oral and IV formations at multiple time points, there was no difference in pain ratings. In another study, rectal paracetamol was shown to have a significant morphine-sparing effect after hysterectomy.

At this time, there has been no study in the gynecologic literature to compare IV to rectal acetaminophen in terms of pain control and effect on overall opioid use in the acute post-operative period.

The rationale for this study is to determine the optimal way of managing post-operative pain in gynecologic surgery in attempt to improve the overall recovery process. More specifically, this study will determine if the route of administration of acetaminophen has an effect on post-operative pain and use of opioid medication following a minimally invasive hysterectomy. The results of this study may guide post-operative pain management after gynecologic surgery, and help limit the amount of opioid use, while potentially reducing pharmacological costs for patients and hospitals.

ELIGIBILITY:
Inclusion Criteria:

* Willing to consent
* Amendable to receive either rectal or intravenous acetaminophen
* Planned hospital stay for at least 24 hours.

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients with a history of regular opioid use prior to surgery based on their current home medication list
* Patients who have required regular opioid intake for the 7 days preceding surgery
* Patients with known hypersensitivity to acetaminophen
* Patients with a baseline preoperative liver function enzymes (AST and ALT) that are greater than twice the upper limits
* Unable to complete procedure as planned.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Aultman Hospital, Canton, Ohio, United States

REFERENCES:
- [Background] Cao X, et al. Effect of intraoperative or postoperative intravenous acetaminophen on postoperative pain scores and opioid requirements in abdominal and spinal surgery patients. Int J Clin Exp Med 11(4)4120-4125, 2018.
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Sconzo Jr FR, Ramamoorthy S. The role of multimodal analgesia in colorectal surgery: a review of clinical data and case-based presentations featuring Ofirmev (acetaminophen) injections. Diseases of the Colon & Rectum 58(2):1-15, 2015.
- [Background] Jibril F, Sharaby S, Mohamed A, Wilby KJ. Intravenous versus Oral Acetaminophen for Pain: Systematic Review of Current Evidence to Support Clinical Decision-Making. Can J Hosp Pharm. 2015 May-Jun;68(3):238-47. doi: 10.4212/cjhp.v68i3.1458. PMID 26157186
- [Background] Petterson PH, Hein A, Owall A, Anderson RE, Jakobsson JG. Early bioavailability in day surgery: a comparison between orally, rectally, and intravenously administered paracetamol. J. of Ambulatory Surgery 12:27-30, 2005.
- [Background] Cobby TF, Crighton IM, Kyriakides K, Hobbs GJ. Rectal paracetamol has a significant morphine-sparing effect after hysterectomy. Br J Anaesth. 1999 Aug;83(2):253-6. doi: 10.1093/bja/83.2.253. PMID 10618939

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Started | 19 | 21
Completed | 17 | 19
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen | Total
Number analyzed (Participants) | 17 | 19 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 17 | 31
  >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.53 (13.64) | 52.37 (14.08) | 51.50 (13.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 17 | 19 | 36
Indication for hysterectomy [Count of Participants; unit: Participants] — Prior to surgery, the indication for surgery was determined based on either clinical (exam based) or histologic findings (tissue biopsy). Based on the clinical and/or histologic findings, patients were scheduled for a hysterectomy for a benign or malignant indication, as determined by the attending physician
  Participants
    Benign | 11 | 12 | 23
    Malignant | 6 | 7 | 13
Diabetes Mellitus [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of diabetes mellitus
  Participants | 4 | 1 | 5
Hypertension [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of hypertension
  Participants | 10 | 7 | 17
Thyroid disease [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of thyroid disease
  Participants | 1 | 2 | 3
Pulmonary disease [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of pulmonary disease
  Participants | 5 | 2 | 7
Anxiety and/or depression [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of anxiety and/or depression
  Participants | 7 | 5 | 12
Obesity [Count of Participants; unit: Participants] — Number of participants with a current diagnosis of obesity (BMI >/= 30)
  Participants | 11 | 14 | 25
Pathology [Count of Participants; unit: Participants] — Based on the microscopic examination of the tissue, the diagnosis of benign or malignant disease was made by a trained pathologist.
  Participants
    Benign | 12 | 13 | 25
    Malignant | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain: Standardized Pain Scale
Description: Post-operative pain control using a standardized pain scale from 0 (no pain) to 10 (worse pain) measured every 4 hours for the 24 hours, or discharge, whichever comes first. Time points were averaged for each participate and reported as a single value.
Time Frame: The first 24 hours following surgery, or upon discharge, whichever comes first.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 19
score on a scale | 2.82 (1.11) | 3.18 (1.26)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = .378, t-test, 2 sided

2. Secondary Outcome: Opioid Use
Description: Total amount of opioid rescue calculated by converting all opiates to Morphine Milligram Equivalents in the first 24 hours following surgery, or upon discharge, whichever comes first.
Time Frame: The first 24 hours following surgery, or upon discharge, whichever comes first.
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 19
Morphine Milligram Equivalents | 25.75 (20.09) | 23.71 (18.46)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = .753, t-test, 2 sided

3. Other Pre Specified Outcome: Postoperative Pain: Standardized Pain Scale
Description: Post-operative pain control using a standardized pain scale from 0 (no pain) to 10 (worse pain) for the first 6 hours after surgery. Time points were averaged for each participate and reported as a single value.
Time Frame: The first 6 hours following surgery
Population: Two participants in the intravenous acetaminophen group were discharged home prior to 6 hours after surgery and therefore were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 17
score on a scale | 3.13 (1.36) | 1.36 (1.78)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.30, t-test, 2 sided

4. Other Pre Specified Outcome: Postoperative Pain: Standardized Pain Scale
Description: Post-operative pain control using a standardized pain scale from 0 (no pain) to 10 (worse pain) for the first 12 hours after surgery. Time points were averaged for each participate and reported as a single value.
Time Frame: The 12 hours following surgery
Population: One participant in the rectal acetaminophen group, and 3 participants in the intravenous acetaminophen group were discharged home prior to 12 hours after surgery and therefore were not included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 16 | 16
score on a scale | 2.99 (1.20) | 3.36 (1.43)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.43, t-test, 2 sided

5. Other Pre Specified Outcome: Opioid Use
Description: Total amount of opioid rescue calculated by converting all opiates to Morphine Milligram Equivalents in the first 6 hours following surgery
Time Frame: The first 6 hours following surgery
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 17
Morphine Milligram Equivalents | 6.74 (7.49) | 7.97 (6.28)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.61, t-test, 2 sided

6. Other Pre Specified Outcome: Opioid Use
Description: Total amount of opioid rescue calculated by converting all opiates to Morphine Milligram Equivalents in the first 12 hours following surgery
Time Frame: The first 12 hours following surgery
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 16 | 16
Morphine Milligram Equivalents | 15.52 (13.35) | 14.17 (11.87)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.77, t-test, 2 sided

7. Other Pre Specified Outcome: Estimated Blood Loss
Description: Total estimated blood loss in millilitres for the surgery
Time Frame: During the duration of the surgery, from start to end time, on average 1.5 hours
Measure: Mean (Standard Deviation); unit: Millilitres
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 19
Millilitres | 273.53 (138.20) | 347.37 (75.41)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.48, t-test, 2 sided

8. Other Pre Specified Outcome: Operative Time
Description: Operative time in minutes determined by the operating room record
Time Frame: From the start to end of the surgery
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
Number analyzed (Participants) | 17 | 19
Minutes | 88.71 (24.22) | 90.89 (21.97)
Statistical Analysis 1: Comparison: Rectal Acetaminophen vs Intravenous Acetaminophen; Test type: Superiority; p = 0.78, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: From administration of acetaminophen until discharge from the hospital, up to 24 hours.
Arm/Group | Rectal Acetaminophen | Intravenous Acetaminophen
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/21
Other Adverse Events (participants affected / at risk) | 0/19 | 0/21

LIMITATIONS AND CAVEATS:
Due to the COVID-19 pandemic, many patients were prohibited to stay overnight in the hospital. Therefore, many patients were discharged home before 24 hours after surgery. This is primarily why the primary and secondary outcomes were analyzed at shorter time intervals (6 hours post-op and 12 hours-op) as well.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT04175509/Prot_SAP_002.pdf
  • Informed Consent Form (2019-10-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT04175509/ICF_001.pdf